CLINICAL TRIAL: NCT02425748
Title: γδ T Cell Immunotherapy for Treatment of
Brief Title: Safety and Efficiency of γδ T Cell Against Non Small Lung Cancer ( Without EGFR Mutation)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Jinan University Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Gd T cell and lung cancer
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2018-06

CONDITIONS: Lung Cancer
Keywords: γδ T Cell, non small lung cancer, Without EGFR Mutation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): DC-CIK cells will be used against tumor cells.
  Interventions: Biological: DC-CIK
- Group B (Experimental): γδ T cells will be used against tumor cells.
  Interventions: Biological: γδ T Cell
- Group C (Experimental): Combination of γδ T cells/ DC-CIK be used against tumor cells.
  Interventions: Biological: γδ T/DC-CIK cells

INTERVENTIONS:
Biological: DC-CIK — DC-CIK cells will be used against tumor cells.
  Arms: Group A
Biological: γδ T Cell — γδ T cells will be used against non small lung tumor.
  Arms: Group B
Biological: γδ T/DC-CIK cells — γδ T/DC-CIK cells will be used against lung tumor.
  Arms: Group C

SUMMARY:
In this study, effects of γδT cells on human non small lung cancer ( without EGFR mutation) in combination with tumor reducing surgery, for example cryosurgery going to be investigated.

DETAILED DESCRIPTION:
Non small lung cancer will be removed using tumor reducing surgery such as cryosurgery. PBMC of the patient will be separated from peripheral blood. After making them potential cancer killer γδ T Cell and DC-CIK, they will be infused to the patients as immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-75
2. Karnofsky performance status >50
3. Diagnosis with non small lung tumors based on histology or the current accepted radiological measures.
4. Classification tumor,nodes,metastasis-classification(TNM) stage: Ⅱ,Ⅲ,Ⅳ Will receive cryosurgery, gd Tcells/ DC-CIK.
5. Life expectancy: Greater than 3 months
6. Ability to understand the study protocol and a willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients with other kinds of cancer
2. History of coagulation disorders or anemia
3. Patients with heart disease and diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Reduced size of the tumor. | Up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China